CLINICAL TRIAL: NCT01512147
Title: Measuring the Effects of Dexmedetomidine on Somatosensory Evoked and Muscular Evoked Potential During Neurosurgery in Pediatric Patients
Brief Title: Dexmedetomidine on Intraoperative Somatosensory and Motor Evoked Potential Monitoring During Neurosurgery in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Heike Gries, MD, PhD, Assistant Professor, Pediatric Anesthesiology, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB00007472
Record Dates: First submitted 2011-12-19; First posted 2012-01-19 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Tethered Spinal Cord; Brain Tumor; Cranio Cervical Compression
Keywords: SSEP measurements; MEP measurements; Pediatric Patients; Neurosurgery; General Anesthesia
MeSH Terms: conditions — Brain Neoplasms | interventions — Isoflurane; Propofol; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Isoflurane, Propofol, Dexmedetomidine (Other): Our trial will examine the changes in latency and amplitude of SSEP and changes in amplitude and morphology of MEP while using different anesthetic combinations including isoflurane, proposal and dexmedetomidine. Monitoring teams will document any changes throughout the surgery and communicate with the team about those changes. The design of the study will be a prospective AB design.
  Interventions: Other: Isoflurane, Propofol, Dexmedetomidine

INTERVENTIONS:
Other: Isoflurane, Propofol, Dexmedetomidine — We will include following general anesthesia techniques:
  Fentanyl 1 - 2 mcg/kg/hr, Propofol 150 - 250 mcg/kg/min, Isoflurane 0.6% expiratory With this general anesthesia technique we will do our first SSEP/MEP measurements after 30 minutes.
  After 30 minutes we will stop isoflurane and will wash out the inhalational anesthetic with high flow air/oxygen and provide:
  Fentanyl 1 - 2 mcg/kg/hr, Propofol 150 - 250mcg/kg/min. This technique will be held for 30 minutes. SSEP/ MEP measurements will be done after 30 minutes.
  After the measurements dexmedetomidine will be added with a loading dose of 0.5 mcg/kg over 10 minutes and continuous infusion of 0.5 mcg/kg/hr for 30 minutes.
  Fentanyl 1 -2 mcg/kg/hr, Propofol 100 - 250mcg/kg/min, Dexmedetomidine 0.5 mcg/kg/hr.

SUMMARY:
The investigators want to know if using the study drug dexmedetomidine will improve nerve wave readings during neurosurgery. These readings are done many times during surgery while the patient is asleep. The readings look at how nerves are working and let the operating team know if nerves are hurt during surgery. If the readings tell that nerves are not working correctly, the surgeons can help while changing the way of operating.

The study drug will be used in addition to the general anesthesia that a patient is given. The nerve readings that the investigators get while using the study drug will be compared with nerve readings that the investigators get while not using the study drug.

The study hypothesis is that dexmedetomidine does not change nerve readings.

DETAILED DESCRIPTION:
Somatosensory evoked potential (SSEP) and motor evoked potential (MEP) have become an integral component in intraoperative care of patients and have resulted in a high degree of sensitivity in predicting neurologic outcomes. According to Padberg, Nuwer and Ecker ,SSEP and MEP monitoring allows surgical interventions to occur early and thus decreases the incidence of postoperative neurologic deficits.

These measurements are done during surgery under general anesthesia and it is known that anesthetic agents have a dose-dependent adverse effect on the ability to record evoked potential responses. All anesthesia agents seem to interfere with the measurements especially in higher doses.

In 1999, dexmedetomidine, a highly specific and selective alpha-2-adrenergic agonist with sedative, anxiolytic and analgesic effects, got FDA approved for adult patients for sedation. Since then, it has also been widely used off-label in various settings; it is described as a successful adjunct for surgical procedures in adolescents and adult populations where SSEP/ MEP monitoring is beneficial. Several small and retrospective studies have shown that dexmedetomidine does not appear to interfere with neurophysiological monitoring when used in FDA approved doses.

In pediatric patients, dexmedetomidine is also used off-label and has been shown to be beneficial. In fact, at Doernbecher Childen's Hospital, the use of dexmedetomidine has become a standard in pediatric procedures involving SSEP and MEP measurements. To the best of our knowledge, prospective studies in pediatric patients with SSEP monitoring while using dexmedetomidine have not been completed.

If dexmedetomidine does not interfere the SSEP/MEP reading, it might be an advantageous adjunct to use in these settings. Propofol has a small risk of a serious side effect called propofol infusion syndrome. Propofol infusion syndrome is potentially life threatening, with the development of a profound lactate acidosis. It is seen when large doses of propofol (usually from a prolonged infusion) are given in the pediatric population.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients between 2 and 12 years old
* Undergoing neurosurgery and
* Requiring SSEP/ MEP measurements

Exclusion Criteria:

* Patients younger than 2 and older than 12 years
* Patients with known bradyarrhythmias
* Patients with severe liver disease
* Conditions that may alter reading, e.g. neuromuscular diseases

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2011-12; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Significant improvement of MEP and SSEP readings during neurosurgery for pediatric patients while using dexmedetomidine as an adjunct to general anesthesia and therefore improvement in clinical decision making. | 30 - 60 minutes of SSEP and MEP measurements intraoperatively
  Changes in latency and amplitude of SSEP and changes in amplitude and morphology of MEP while using different anesthetic combinations including isoflurane, propofol and dexmedetomidine.

CONTACTS AND LOCATIONS:
Overall Officials: Heike Gries, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Ohsu - Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- [Background] Padberg AM, Wilson-Holden TJ, Lenke LG, Bridwell KH. Somatosensory- and motor-evoked potential monitoring without a wake-up test during idiopathic scoliosis surgery. An accepted standard of care. Spine (Phila Pa 1976). 1998 Jun 15;23(12):1392-400. doi: 10.1097/00007632-199806150-00018. PMID 9654631
- [Background] Ecker ML, Dormans JP, Schwartz DM, Drummond DS, Bulman WA. Efficacy of spinal cord monitoring in scoliosis surgery in patients with cerebral palsy. J Spinal Disord. 1996 Apr;9(2):159-64. PMID 8793785
- [Background] Nuwer MR, Dawson EG, Carlson LG, Kanim LE, Sherman JE. Somatosensory evoked potential spinal cord monitoring reduces neurologic deficits after scoliosis surgery: results of a large multicenter survey. Electroencephalogr Clin Neurophysiol. 1995 Jan;96(1):6-11. doi: 10.1016/0013-4694(94)00235-d. PMID 7530190
- [Background] Thuet ED, Padberg AM, Raynor BL, Bridwell KH, Riew KD, Taylor BA, Lenke LG. Increased risk of postoperative neurologic deficit for spinal surgery patients with unobtainable intraoperative evoked potential data. Spine (Phila Pa 1976). 2005 Sep 15;30(18):2094-103. doi: 10.1097/01.brs.0000178845.61747.6a. PMID 16166902
- [Background] Banoub M, Tetzlaff JE, Schubert A. Pharmacologic and physiologic influences affecting sensory evoked potentials: implications for perioperative monitoring. Anesthesiology. 2003 Sep;99(3):716-37. doi: 10.1097/00000542-200309000-00029. No abstract available. PMID 12960558
- [Background] Bhana N, Goa KL, McClellan KJ. Dexmedetomidine. Drugs. 2000 Feb;59(2):263-8; discussion 269-70. doi: 10.2165/00003495-200059020-00012. PMID 10730549
- [Background] Tobias JD, Goble TJ, Bates G, Anderson JT, Hoernschemeyer DG. Effects of dexmedetomidine on intraoperative motor and somatosensory evoked potential monitoring during spinal surgery in adolescents. Paediatr Anaesth. 2008 Nov;18(11):1082-8. doi: 10.1111/j.1460-9592.2008.02733.x. PMID 18717802
- [Background] Bala E, Sessler DI, Nair DR, McLain R, Dalton JE, Farag E. Motor and somatosensory evoked potentials are well maintained in patients given dexmedetomidine during spine surgery. Anesthesiology. 2008 Sep;109(3):417-25. doi: 10.1097/ALN.0b013e318182a467. PMID 18719439
- [Background] Anschel DJ, Aherne A, Soto RG, Carrion W, Hoegerl C, Nori P, Seidman PA. Successful intraoperative spinal cord monitoring during scoliosis surgery using a total intravenous anesthetic regimen including dexmedetomidine. J Clin Neurophysiol. 2008 Feb;25(1):56-61. doi: 10.1097/WNP.0b013e318163cca6. PMID 18303561
- [Background] Mahmoud M, Sadhasivam S, Salisbury S, Nick TG, Schnell B, Sestokas AK, Wiggins C, Samuels P, Kabalin T, McAuliffe J. Susceptibility of transcranial electric motor-evoked potentials to varying targeted blood levels of dexmedetomidine during spine surgery. Anesthesiology. 2010 Jun;112(6):1364-73. doi: 10.1097/ALN.0b013e3181d74f55. PMID 20460997
- [Background] Bloom M, Beric A, Bekker A. Dexmedetomidine infusion and somatosensory evoked potentials. J Neurosurg Anesthesiol. 2001 Oct;13(4):320-2. doi: 10.1097/00008506-200110000-00007. PMID 11733664
- [Background] Moller AR. Intraoperative neurophysiologic monitoring. Am J Otol. 1995 Jan;16(1):115-7. No abstract available. PMID 8579167